CLINICAL TRIAL: NCT07029490
Title: Enhancing Mammography Programs for Outreach, Wellness, Education, and Resources (EMPOWER) in Underserved Populations Study
Acronym: EMPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HCI185522; SPA-RFA-Team23-1001996-01-PASD (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Mammography; Chatbot; Mobile Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual Care: This will include participants randomized to usual care.
- Chatbot (Experimental): Chatbot: This will include participants randomized to usual care with the Chatbot.
  Interventions: Other: Chatbot

INTERVENTIONS:
Other: Chatbot — The Chatbot used in this study will be used after mammography to facilitate follow-up, answer patient questions, and provide information.
  Arms: Chatbot

SUMMARY:
This study is investigating the feasibility of a digital tool called a chatbot for providing educational information about mammography through a tablet, computer, or phone. This study will recruit participants who recently had a mammogram with the University of Utah. Based on their mammography results, women will be placed into two cohorts using their BI-RADS category. Once mammogram results are available, patients will be randomized 1:1 to either usual care or usual care with chatbot. This study will randomly invite participants from four groups for focus group discussions (FGDs) based on their mammogram results and adherence to screening recommendations

DETAILED DESCRIPTION:
Breast cancer screening inequities are drivers of disparities for rural and Latina women.

Chatbots are increasingly popular in various healthcare contexts and can be easily accessed through smartphones, tablets, laptops, and desktops. Chatbots have many advantages for patient messaging, including providing scripted education and motivational information interactively, chunking information into digestible segments, and allowing for choice in the amount of information received at any one time. Thus, with chatbots this study can tailor the interaction based on individual patient factors. Chatbots are accessible to the vast majority of U.S. adults. While chatbots have been used successfully in some clinical contexts, there is a lack of studies that investigated the use of chatbots as part of a mobile screening program to increase adherence to follow-up recommendations about either screening or diagnostic care.

Study staff will approach women at the time of or soon after a patient's routine breast cancer screening and invite the patient to participate in the study. Participants will complete baseline surveys at time of enrollment. This survey includes demographics and preferred contact method (e.g., text, email) that will be used to initiate the chatbot communication which can be completed via phone or website. Usual clinical procedures will be used to interpret participants' routine screening mammograms, including the use of the breast imaging-reporting and data system (BI-RADS), typically within 1 week of imaging.

Based on their mammography results, women will be placed into two cohorts using their BI-RADS category.

All participants will complete follow-up questionnaires, available in English and Spanish. For the follow-up surveys, the research team will contact participants via their preferred method (text or email) and send a link to the follow-up survey. If unsuccessful, the research team will then contact participants by phone to complete the survey via text or call.

Once mammogram results are available, patients will be randomized 1:1 to either usual care or usual care with chatbot, with randomization in permuted blocks of size and stratified by age (<55 vs. ≥55 years, a proxy for menopause and indicator of risk); rural/frontier vs. urban; language preference (English vs. Spanish); and cohort (normal vs. abnormal result).

This study will randomly invite participants from four groups for focus group discussions (FGDs) based on their mammogram results and adherence to screening recommendations. This study aim to conduct 8 FGDs (2 per group, one in Spanish and one in English) with 8-10 participants each.

ELIGIBILITY:
Inclusion Criteria:

* Adult (equal to or above 18 years old)
* English or Spanish speaking
* Visit a mammography program for routine screening.

Exclusion Criteria:

* Patients who are currently in treatment for breast cancer
* Patients who are not of 18 years of age.
* Patients who don't speak English or Spanish
* Men
* Cognitive limitations that impede informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2700 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Screening Adherence | up to 24 months from initiation of study intervention
  This outcome measure will test the addition of virtual navigation to usual processes of care to increase screening adherence for underserved women undergoing mobile mammography who have an abnormal breast cancer screening exam.
  Screening adherence will be measured as a two-point survey item (Yes/No). This outcome measure will report the proportion of participants who self-reported screening adherence.

SECONDARY OUTCOMES:
Receipt of follow-up testing | up to 12 months from initiation of study intervention
  This outcome measure will test the addition of virtual navigation to usual processes of care to increase follow-up testing for underserved women undergoing mobile mammography who have an abnormal breast cancer screening exam.
  Receipt of follow-up testing will be measured as survey items. For subjects who were recommended to have additional breast imaging or a breast biopsy, this will report if they completed the recommendation.
  This outcome measure will report the proportion of individuals who received all recommended follow-up tests after an initial breast screening indicating additional breast imaging or biopsy.
Receipt of episode completion | up to 12 months from initiation of study intervention
  This outcome measure will test the addition of virtual navigation to usual processes of care to increase episode completion for underserved women undergoing mobile mammography who have an abnormal breast cancer screening exam.
  Receipt of episode completion will be measured through a survey. This outcome measure will report the proportion of subjects who complete all recommended follow-up steps after initial breast cancer screening or diagnosis, including imaging, biopsy, specialist appointments, and initiation of treatment if applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute/ University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer Stat Facts: Female Breast Cancer. https://seer.cancer.gov/statfacts/html/breast.html. Accessed Oct 11, 2021.
- [Background] American Cancer Society. Cancer Facts & Figures for Hispancis/Latinos 2018-2020. Atlanta: American Cancer Society, Inc.;2018.
- [Background] Death Rates for Selected Cancers by Race and Ethnicity, US, 2010-2014. 2016; https://www.cancer.org/content/dam/cancer-org/research/cancer-facts-and-statistics/annual-cancer-facts-and-figures/2017/death-rates-for-selected-cancers-by-race-and-ethnicity-us-2010-2014.pdf. Accessed Oct 11, 2021.
- [Background] Henry KA, Sherman R, Farber S, Cockburn M, Goldberg DW, Stroup AM. The joint effects of census tract poverty and geographic access on late-stage breast cancer diagnosis in 10 US States. Health Place. 2013 May;21:110-21. doi: 10.1016/j.healthplace.2013.01.007. Epub 2013 Mar 1. PMID 23454732
- [Background] DeSantis CE, Ma J, Goding Sauer A, Newman LA, Jemal A. Breast cancer statistics, 2017, racial disparity in mortality by state. CA Cancer J Clin. 2017 Nov;67(6):439-448. doi: 10.3322/caac.21412. Epub 2017 Oct 3. PMID 28972651
- [Background] Doescher MP, Jackson JE. Trends in cervical and breast cancer screening practices among women in rural and urban areas of the United States. J Public Health Manag Pract. 2009 May-Jun;15(3):200-9. doi: 10.1097/PHH.0b013e3181a117da. PMID 19363399
- [Background] Roche LM, Niu X, Stroup AM, Henry KA. Disparities in Female Breast Cancer Stage at Diagnosis in New Jersey: A Spatial-Temporal Analysis. J Public Health Manag Pract. 2017 Sep/Oct;23(5):477-486. doi: 10.1097/PHH.0000000000000524. PMID 28430705
- [Background] Williams F, Jeanetta S, O'Brien DJ, Fresen JL. Rural-urban difference in female breast cancer diagnosis in Missouri. Rural Remote Health. 2015 Jul-Sep;15(3):3063. Epub 2015 Jul 29. PMID 26223824
- [Background] Bennett KJ, Pumkam C, Bellinger JD, Probst JC. Cancer screening delivery in persistent poverty rural counties. J Prim Care Community Health. 2011 Oct 1;2(4):240-9. doi: 10.1177/2150131911406123. Epub 2011 May 17. PMID 23804842
- [Background] Bennett KJ, Probst JC, Bellinger JD. Receipt of cancer screening services: surprising results for some rural minorities. J Rural Health. 2012 Jan;28(1):63-72. doi: 10.1111/j.1748-0361.2011.00365.x. Epub 2011 Mar 11. PMID 22236316
- [Background] Coughlin SS, Leadbetter S, Richards T, Sabatino SA. Contextual analysis of breast and cervical cancer screening and factors associated with health care access among United States women, 2002. Soc Sci Med. 2008 Jan;66(2):260-75. doi: 10.1016/j.socscimed.2007.09.009. Epub 2007 Nov 19. PMID 18022299
- [Background] Horner-Johnson W, Dobbertin K, Iezzoni LI. Disparities in receipt of breast and cervical cancer screening for rural women age 18 to 64 with disabilities. Womens Health Issues. 2015 May-Jun;25(3):246-53. doi: 10.1016/j.whi.2015.02.004. Epub 2015 Apr 9. PMID 25864023
- [Background] Leung J, McKenzie S, Martin J, McLaughlin D. Effect of rurality on screening for breast cancer: a systematic review and meta-analysis comparing mammography. Rural Remote Health. 2014;14(2):2730. Epub 2014 Jun 23. PMID 24953122
- [Background] Incidence Rates for Utah by County Breast (Late Stage), 2014-2018, All Races (includes Hispanic), Female, All Ages. https://statecancerprofiles.cancer.gov/map/map.withimage.php?49&county&001&055211&00&2&11&0&1&5&0#results. Accessed Oct 11, 2021.
- [Background] Guillaume E, Launay L, Dejardin O, Bouvier V, Guittet L, Dean P, Notari A, De Mil R, Launoy G. Could mobile mammography reduce social and geographic inequalities in breast cancer screening participation? Prev Med. 2017 Jul;100:84-88. doi: 10.1016/j.ypmed.2017.04.006. Epub 2017 Apr 10. PMID 28408217